CLINICAL TRIAL: NCT03298334
Title: Vaginal Microbiome Seeding and Health Outcomes in Cesarean-delivered Neonates: a Randomized Controlled Trial
Brief Title: Vaginal Microbiome Seeding and Health Outcomes in Cesarean-delivered Neonates.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins University (Other); Rutgers University (Other); Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-2694
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Cesarean Delivery Affecting Newborn; Obesity, Childhood; Intestinal Microbiome; Microbiota; Host Microbial Interactions; Gastrointestinal Microbiome
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Receives Vaginal Seeding (Active Comparator)
  Interventions: Biological: Vaginal Seeding
- No Vaginal Seeding (Sham Comparator)
  Interventions: Other: No Vaginal Seeding

INTERVENTIONS:
Biological: Vaginal Seeding — A gauze containing the Mother's vaginal flora will be swabbed over the face and body of the neonate shortly after cesarean delivery.
  Arms: Receives Vaginal Seeding
Other: No Vaginal Seeding — A gauze carrying sterile saline will be swabbed over the face and body of the neonate shortly after cesarean delivery.
  Arms: No Vaginal Seeding

SUMMARY:
Neonates delivered by scheduled Cesarean Section will be randomized to receive vaginal seeding (exposing the infant to Mother's vaginal flora) or sham. Infants will be followed for three years to examine health outcomes including microbiome development, immune development, metabolic outcomes, and any adverse events.

DETAILED DESCRIPTION:
Cesarean section (CS) delivery is a common surgical procedure intended to increase the chances of successful delivery and to protect the health of the mother and baby. Yet this intervention is overused and has been associated with higher risk of immune and metabolic disorders in the offspring. It is hypothesized that these associations are due to CS-delivered newborns not receiving the full inoculum of maternal microbes at birth.

While restoring labor is not possible, restoring the microbes that colonize infants during birth through exposure to vaginal flora, is feasible, and has been shown in a small pilot study, to normalize the microbiota of the intestine, skin and mouth during the first month of life.

The investigators hypothesize that the restoration of the vaginal microbiota to the infant at birth will restore the infant microbiome and decrease the risk of obesity and other immune-mediated diseases linked with CS. The investigators aim to test this hypothesis in a randomized controlled trial by first examining the effect of vaginal seeding, in CS-delivered newborns, on the gut microbiota composition, structure and function (Phase I of study; first 50 infants) and then on the BMI z score and other immune-mediated outcomes (Phase II of study; 600 infants).

Methods: CS-delivered neonates will be randomized to either an experimental arm with exposure to the maternal vaginal microbiota at birth, or a control arm with no exposure. Feces, skin, saliva, breast milk, and vaginal swabs will be collected for microbiome analysis. The investigators will obtain clinical information from in-person visits, surveys and the electronic health record.

Implications: this randomized controlled clinical study will provide evidence of whether the "vaginal seeding" procedure can safely transfer microbes from mom-to-baby, and whether these microbes are beneficial for the metabolic and immune health of the child.

ELIGIBILITY:
Inclusion Criteria for Mother:

* Scheduled for cesarean delivery at ≥ 37 weeks
* Pregnant with single fetus, in good general health, age 18 years or older
* Negative maternal testing for infections transmitted through vaginal and/or other body fluids performed as standard of care tests in early pregnancy
* Negative testing for Group B strep at 35-37 weeks gestation
* Vaginal pH ≤ 4.5 indicative of Lactobacillus-dominated vaginal microbiota
* No maternal or fetal complications that may inhibit the ability to perform microbiome restoration per protocol
* English or Spanish speaking
* Negative maternal testing for Gonorrhea, Chlamydia, Hepatitis B, Hepatitis C, Syphilis, and HIV at 35 weeks gestation or later
* Women aged 18-29 years must have a normal Pap test within 3 years
* Women aged 30-65 years must have a normal Pap test and an HPV test (co-testing) within 5 years or FDA-approved primary hrHPV testing alone within 5 years or a normal Pap test alone within 3 years
* Negative maternal testing for SARS-CoV-2 for the delivery admission performed as standard of care test at the Inova Health System.

Inclusion Criteria for Infant:

* Infant condition after delivery requires no more than standard neonatal resuscitation* or is otherwise medically unable to receive the full VMT procedure

[*] Standard neonatal resuscitation may include: tactile stimulation, bulb suction, oxygen without positive pressure, or drying

Exclusion Criteria for Mother:

* Delivery at a hospital other than Inova Health System
* Cesarean delivery scheduled for active infection that would have interfered with vaginal delivery such as genital herpetic lesions
* Rupture of membranes prior to scheduled cesarean delivery
* Bacterial vaginosis within 30 days of cesarean delivery
* Symptomatic urinary tract infection within 30 days of cesarean delivery
* Antibiotic therapy within 30 days of cesarean delivery (exclusive of medication use for prophylaxis at the time of surgery)
* Symptoms on admission suggesting Chorioamnionitis, e.g. maternal fever, fundal tenderness
* Symptoms on delivery admission of possible vaginal infection such as genital herpetic lesions
* History of genital HSV
* History positive testing for Group B strep infection
* History of a child with a diagnosis of Group B strep sepsis
* Pregnancy a result of donor egg or surrogacy
* Preexisting history of Type I or Type II Diabetes
* Maternal history of documented genital HPV infection, positive HPV testing or genital warts on physician examination
* Positive maternal testing for SARS-CoV-2 within 30 days of delivery or symptoms on admission suggesting potential Covid-19 infection

Ages: 0 Days to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Adiposity | 2 years
  E.g. Body mass index z-score

SECONDARY OUTCOMES:
Adverse events | 3 years
  Monitoring for adverse events
Intestinal microbiota | 3 years
  Intestinal microbiota development over the first three years of life
Immune and inflammatory regulation | 3 years
  E.g. Monitoring for immune and inflammatory mediated conditions

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Hourigan, MD, Chief, Clinical Microbiome Unit, NIAID, Pediatric Gastroenterologist, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID), Inova Children's Hospital; Noel Mueller, PhD, Principal Investigator — Johns Hopkins University; Maria Gloria Dominguez Bello, PhD, Principal Investigator — Rutgers University; Lawrence Appel, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Inova Health System, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared with co-principal investigators (Maria Gloria Dominguez-Bello at Rutgers University and Noel Mueller at Johns Hopkins School of Medicine).
Supporting Information: Study Protocol, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Dominguez-Bello MG, De Jesus-Laboy KM, Shen N, Cox LM, Amir A, Gonzalez A, Bokulich NA, Song SJ, Hoashi M, Rivera-Vinas JI, Mendez K, Knight R, Clemente JC. Partial restoration of the microbiota of cesarean-born infants via vaginal microbial transfer. Nat Med. 2016 Mar;22(3):250-3. doi: 10.1038/nm.4039. Epub 2016 Feb 1. PMID 26828196
- [Background] Song SJ, Wang J, Martino C, Jiang L, Thompson WK, Shenhav L, McDonald D, Marotz C, Harris PR, Hernandez CD, Henderson N, Ackley E, Nardella D, Gillihan C, Montacuti V, Schweizer W, Jay M, Combellick J, Sun H, Garcia-Mantrana I, Gil Raga F, Collado MC, Rivera-Vinas JI, Campos-Rivera M, Ruiz-Calderon JF, Knight R, Dominguez-Bello MG. Naturalization of the microbiota developmental trajectory of Cesarean-born neonates after vaginal seeding. Med. 2021 Aug 13;2(8):951-964.e5. doi: 10.1016/j.medj.2021.05.003. Epub 2021 Jun 17. PMID 35590169
- [Background] Hourigan SK, Dominguez-Bello MG, Mueller NT. Can maternal-child microbial seeding interventions improve the health of infants delivered by Cesarean section? Cell Host Microbe. 2022 May 11;30(5):607-611. doi: 10.1016/j.chom.2022.02.014. PMID 35550663
- [Derived] Namasivayam S, Tilves C, Ding H, Wu S, Domingue JC, Ruiz-Bedoya C, Shah A, Bohrnsen E, Schwarz B, Bacorn M, Chen Q, Levy S, Dominguez Bello MG, Jain SK, Sears CL, Mueller NT, Hourigan SK. Fecal transplant from vaginally seeded infants decreases intraabdominal adiposity in mice. Gut Microbes. 2024 Jan-Dec;16(1):2353394. doi: 10.1080/19490976.2024.2353394. Epub 2024 May 14. PMID 38743047